CLINICAL TRIAL: NCT00690222
Title: A Comparison of Intracameral Phenylephrine 2% and Tropicamide 0.2% With Topical Phenylephrine 2.5% and Tropicamide 1% for Pupillary Dilation During Cataract Surgery on Patients With and Without Pseudoexfoliation Syndrome.
Brief Title: Intracameral Mydriasis Versus Topical Mydriasis in Cataract Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHDA-RS/2008-024
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2008-05

CONDITIONS: Cataract; Phacoemulsification; Mydriasis; Pseudoexfoliation Syndrome
Keywords: cataract surgery; phacoemulsification; pupil; dilation; mydriasis; intracameral; topical; pseudoexfoliation syndrome
MeSH Terms: conditions — Cataract; Mydriasis; Exfoliation Syndrome; Dilatation, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- TM (No Intervention): Topical mydriasis without pseudoexfoliation
- ICM (Experimental): Intracameral mydriasis without pseudoexfoliation
  Interventions: Procedure: Intracameral injection of mydriatic agent
- TM - PXF (No Intervention): Topical mydriasis with pseudoexfoliation
- ICM - PXF (Experimental): Intracameral Mydriasis with pseudoexfoliation
  Interventions: Procedure: Intracameral injection of mydriatic agent

INTERVENTIONS:
Procedure: Intracameral injection of mydriatic agent — A mixture of 0.2 % tropicamide and 2% phenylephrine will be injected into the anterior chamber at the beginning of surgery
  Arms: ICM; ICM - PXF

SUMMARY:
The purpose is to determine if an intracameral solution of 0.2% tropicamide and 2% phenylephrine can dilate the pupil for cataract surgery as well as pre-operative topical 1% tropicamide and 5% phenylephrine. We will be looking at two separate groups of patients, those with and those without pseudoexfoliation syndrome.

We will be looking at how each method affects the size of the pupil at the beginning and at the end of cataract surgery. In addittion, we will look at what effect the two different methods have on blood pressure and heart rate in the pre-operative, peri-operative and post-operative periods.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give consent
* Greater than 18 years of age
* Planned clear cornea cataract extraction and placement of foldable posterior chamber intraocular lens
* No secondary procedure planned (i.e. trabeculectomy, keratectomy, corneal transplant, vitreo-retinal procedure etc.)
* Systemic condition capable of undergoing topical anesthesia
* No previous intraocular surgery
* Pseudoexfoliation syndrome (PXF) for group 1
* No Pseudoexfoliation syndrome for group 2

Exclusion Criteria:

* Not fulfilling inclusion criteria
* Any iris pathology including but not limited to posterior synechia, iridocorneal endothelial syndrome, corectopia, traumatic mydriasis, Horner's syndrome, Adie's pupil, cyclodialysis, iridodialysis
* Previous or concurrent use of Flomax® or similar alpha-antagonist medication
* Corneal pathology affecting pupil magnification or measurement (keratoconus, peripheral thinning, sclerocornea, scarring)
* Uncontrolled Hypertension (greater than 170/90 on pre-operative assessment on day of surgery as measured by automated DATEX monitor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pupil size | At beginning and completion of cataract surgery

SECONDARY OUTCOMES:
Blood pressure | Peri-operatively
Heart rate | Peri-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada